CLINICAL TRIAL: NCT04673409
Title: Multiparametric Tissue Characterisation of Myocardial Inflammation in Autoimmune Rheumatic Diseases (AIRD) Using Cardiovascular Magnetic Resonance Imaging
Brief Title: CMR Imaging of Autoimmune Diseases
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 258879; 20/L0/1076 (Other: Research Ethics Committee (United Kingdom))
Record Dates: First submitted 2020-11-30; First posted 2020-12-17 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2023-10

CONDITIONS: Myocarditis; Autoimmune Rheumatologic Disease
Keywords: Cardiovascular Magnetic Resonance Imaging; Inflammation
MeSH Terms: conditions — Myocarditis; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Suspected myocarditis of undefined aetiology: Patients with signs and symptoms of acute myocarditis (as defined by the European Society of Cardiology Working Group on Myocardial and Pericardial Diseases).
  Interventions: Diagnostic Test: Novel Cardiac MRI sequences
- Suspected myocarditis with autoimmune rheumatic disease: Patients with suspected myocarditis due to an underlying AIRD.
  Interventions: Diagnostic Test: Novel Cardiac MRI sequences

INTERVENTIONS:
Diagnostic Test: Novel Cardiac MRI sequences — Novel CMR sequences that allow accurate multiparametric evaluation of the whole myocardium with 3D high spatial resolution and in a patient-friendly free-breathing approach in a predictable amount of scanning time (3D T2 mapping and 3D anatomical and LGE imaging). This will be compared to the data acquired with conventional/2D sequences.

SUMMARY:
Myocarditis is an important clinical problem which can can occur as a result of viral infections and autoimmune rheumatic diseases. Cardiac MRI is an important non-invasive means of making a diagnosis. However, current MRI techniques have significant limitations. Firstly, in order to create high-quality pictures, patients are required to hold their breath several times for multiple lengths of time. They often struggle with this due to underlying heart/lung problems. This can adversely affect the overall quality and image interpretation. Secondly, current techniques create 2D images that are potentially underestimating the presence and severity of any tissue inflammation/ injury. This may result in inappropriate treatment, particularly for patients with underlying autoimmune systemic disease who require immunosuppression.

Diagnosis by MRI rests on detecting tissue injury through T2 and T1-weighted sequences which detect tissue inflammation and tissue injury. The purpose of this study is to evaluate the diagnostic accuracy of novel 3D free-breathing sequences for T2-weighted and fibrosis/ LGE imaging.

Patients with suspected isolated myocarditis (viral/idiopathic) or myocarditis as part of an autoimmune systemic disease will be recruited to ensure that the novel techniques are tested in a broad spectrum of patients with inflammatory heart muscle disease.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for CMR for clinically suspected myocarditis either idiopathic or in the context of autoimmune rheumatic disease.
* Patients who are able to give informed consent.

Exclusion Criteria:

* Patients in atrial fibrillation.
* Patients who are unable to give informed consent.
* Patients whose physical or mental condition indicates that the additional time in the CMR scanner should be minimised.
* Patients who cannot have CMR due to either contraindications to CMR (e.g., non-conditional intracardiac devices) or contraindications to contrast (e.g., history of allergy to gadolinium).

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the acute cardiology service and the rheumatology service referred for cardiovascular magnetic resonance imaging.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of novel versus conventional sequences | 2 weeks
  The CMR diagnosis of myocarditis will be made according to the revised (2018) Lake Louise criteria which mandate an increase in T2 (signal intensity in arbitrary units or absolute values in ms) and a T1-based marker (either absolute T1 in ms or LGE). T2-times and LGE from the novel 3D sequences will be combined as per revised Lake Louise criteria recommendations to make a diagnosis and compared with the conventional clinical sequences. A clinical diagnosis of cardiovascular inflammation will be made by an expert consensus adjudication panel initially based on evaluation of the patient's history and examination findings; ECG; the results of laboratory testing; and ancillary imaging findings. To avoid incorporation bias, the initial assessment will be blinded to tissue characterisation findings, and the classification will be compared between new and old methods using ROC analysis and the DeLong test.

SECONDARY OUTCOMES:
Quantitative accuracy and precision of novel 3D sequences compared with conventional sequences | 2 weeks
  The accuracy (bias) and precision (95% limits of agreement) of the novel 3D quantitative T2-mapping sequence will be assessed with the conventional 2D-values as a reference comparator using the methods of Bland and Altman. This will be used to derive the bias in measured T2 times in ms and the corresponding 95% limits of agreement (in ms).
Acquisition time for both conventional and novel sequences versus conventional sequences | 2 weeks
Proportion of diagnostic images with novel versus conventional sequences | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tevfik F. Ismail, PhD, FSCMR, Principal Investigator — King's College London
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No